CLINICAL TRIAL: NCT01054547
Title: Local Anesthetic Activity of Liposomal Formulations in Dentistry
Brief Title: Topical Formulations of Liposomal Local Anesthetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Michelle Franz-Montan, Unicamp
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 093/2006
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2006-05

CONDITIONS: Administration, Topical Drug; Administration, Topical; Anesthetic Drugs
Keywords: topical anesthetic; liposomal ropivacaine; dentistry
MeSH Terms: interventions — Ropivacaine; Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal ropivacaine, topical (Placebo Comparator): The topical anesthetics were applied at the region of right and left maxillary lateral incisors at the buccal mucosa.
  Interventions: Drug: Ropivacaine
- Liposomal ropivacaine, palatal mucosa (Placebo Comparator): Topical formulations were applied at the palatal mucosa at the right canine region and efficacy of topical formulations was accessed through insertion of a 30 gauge needle and injection of anesthetic solution.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 100 mg of the following formulations: Liposome-encapsulated 1 and 2% ropivacaine gel, liposome placebo gel and 2.5% lidocaine and 2.5% prilocaine cream were applied once during 5 minutes.
  Other Names: Topical anesthesia in the palatal mucosa
  Arms: Liposomal ropivacaine, palatal mucosa
Drug: Ropivacaine — 100 mg of the following formulations: Liposome-encapsulated 1 and 2% ropivacaine gel, liposome placebo gel and 20% benzocaine gel were applied once during 30 minutes.
  Other Names: Topical anesthesia in the buccal mucosa.
  Arms: Liposomal ropivacaine, topical

SUMMARY:
This blinded cross-over study aim to evaluate the efficacy of topical liposome-encapsulated ropivacaine formulations.

DETAILED DESCRIPTION:
This blinded cross-over study aim to evaluate the efficacy of topical liposome-encapsulated 1 and 2% ropivacaine gel formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders and allergy to local anesthetics

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
After topical application of the local anesthetic formulations at the oral mucosa, their influence on pulpal response was assessed by an electrical pulp tester. | 10 minutes

SECONDARY OUTCOMES:
The efficacy of the topical anesthetics was measured after a simulation of a local anesthesia in the application site (insertion of a 30 gauge needle until periosteum contact). | 10 seconds after removal of topical formulation

CONTACTS AND LOCATIONS:
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Franz-Montan M, de Paula E, Groppo FC, Silva AL, Ranali J, Volpato MC. Liposome-encapsulated ropivacaine for intraoral topical anesthesia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Dec;110(6):800-4. doi: 10.1016/j.tripleo.2010.07.005. PMID 21112538
- [Derived] Franz-Montan M, de Paula E, Groppo FC, Silva AL, Ranali J, Volpato MC. Liposomal delivery system for topical anaesthesia of the palatal mucosa. Br J Oral Maxillofac Surg. 2012 Jan;50(1):60-4. doi: 10.1016/j.bjoms.2010.10.018. Epub 2010 Nov 23. PMID 21106282